CLINICAL TRIAL: NCT00340275
Title: Longitudinal Study of Vaginal Flora
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999023; OH99-CH-N023
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-18

CONDITIONS: Vaginal Flora
Keywords: Bacterial Vaginosis; Vaginal Infection; Vaginitis; Cohort Study; Sexually Transmitted Disease
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis; Sexually Transmitted Diseases

SUMMARY:
Bacterial vaginosis is a syndrome manifested by adverse alterations in vaginal microbial flora. It is present in 10 to 25% of women in the general population, and is the most common vaginal infection. It has been associated with a number of adverse sequelae in reproductive health including acquisition of HIV, pelvic inflammatory disease, cervical dysplasia, and complications of gynecological procedures. During pregnancy it has been associated with an increased risk of preterm birth an postpartum maternal infection. However, the vaginal microbial flora remains poorly understood. Information on variation in microbial flora and its association with BV from a longitudinal study is unavailable. This prospective observational study aims to advance our knowledge of the natural history and abnormal alteration in vaginal microbial flora, and to identify risk factors that are associated with these changes. A total of 5500 healthy, non-pregnant women of reproductive age will be enrolled and followed up in Birmingham, Alabama, for one year (baseline visit plus once every three months afterwards, totaling 5 visits). Detailed information on sociodemographic status, medical history, hygiene practice, sexual behavior and psychosocial stress will be collected through in-person interviews. Routine gynecological and dental examinations will be carried out during the study visits. Samples of vaginal secretion and blood will be collected. Laboratory tests to quantify vaginal microbial flora and to identify infection of bacterial vaginosis as well as common sexually transmitted diseases will be conducted. This project is expected to complete in 5 years.

DETAILED DESCRIPTION:
Bacterial vaginosis is a syndrome manifested by adverse alterations in vaginal microbial flora. It is present in 10 to 25% of women in the general population, and is the most common vaginal infection. It has been associated with a number of adverse sequelae in reproductive health including acquisition of HIV, pelvic inflammatory disease, cervical dysplasia, and complications of gynecological procedures. During pregnancy it has been associated with an increased risk of preterm birth and postpartum maternal infection. However, the vaginal microbial flora remains poorly understood. Information on variation in microbial flora and its association with BV from a longitudinal study is unavailable. This prospective observational study aims to advance our knowledge of the natural history and abnormal alteration in vaginal microbial flora, and to identify risk factors that are associated with these changes. A total of 5500 healthy, non-pregnant women of reproductive age will be enrolled and followed up in Birmingham, Alabama, for one year (baseline visit plus once every three months afterwards, totaling 5 visits). Detailed information on sociodemographic status, medical history, hygiene practice, sexual behavior and psychosocial stress will be collected through in-person interviews. Routine gynecological and dental examinations will be carried out during the study visits. Samples of vaginal secretion and blood will be collected. Laboratory tests to quantify vaginal microbial flora and to identify infection of bacterial vaginosis as well as common sexually transmitted diseases will be conducted. This project is expected to complete in 5 years.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Females, age 15-44.
* Since bacterial vaginosis is primarily a condition of reproductive-age women, this study will be restricted to women regarded by demographers as reproductive age.
* Non-pregnant women whose last menstrual period is later than expected will undergo a urine pregnancy test. Women who become pregnant while on study will complete their next regularly scheduled study visit, following which their participation will terminate.

EXCLUSION CRITERIA:

1. Immunocompromised status

   Receiving or expected to receive in the next 12 months cytotoxic or immunosuppressive drugs.

   Receiving or expected to receive in the next 12 months one or more 30-day courses of corticosteroids.

   Congenital or acquired immune deficiency; known HIV positivity.
2. Primary or secondary affective disorder, psychosis, emotional or intellectual limitations that preclude informed consent.
3. Non-fluency in English.
4. Post-menopausal (natural or surgical).
5. Status post hysterectomy or expected to undergo hysterectomy in the next 12 months.
6. Status post pelvic radiotherapy, or expected to undergo pelvic radiotherapy in the next 12 months.
7. Receiving or expected to receive chronic (daily for at least 30 days) antibiotics in the next 12 months.
8. Planning to move out of the area in the next 12 months.
9. Participating or expected to participate during the next 12 months in a clinical trial in which antibiotics or topical microbicides will be administered in a blinded manner.
10. Women who unexpectedly develop one of these conditions during their participation will continue to be followed, unless a specific contraindication arises.

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5500 (Estimated)
Dates: Start 1999-04-14; Study Completion 2010-11-18

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Background] Goldenberg RL, Klebanoff MA, Nugent R, Krohn MA, Hillier S, Andrews WW. Bacterial colonization of the vagina during pregnancy in four ethnic groups. Vaginal Infections and Prematurity Study Group. Am J Obstet Gynecol. 1996 May;174(5):1618-21. doi: 10.1016/s0002-9378(96)70617-8. PMID 9065140
- [Background] Amsel R, Totten PA, Spiegel CA, Chen KC, Eschenbach D, Holmes KK. Nonspecific vaginitis. Diagnostic criteria and microbial and epidemiologic associations. Am J Med. 1983 Jan;74(1):14-22. doi: 10.1016/0002-9343(83)91112-9. PMID 6600371
- [Background] Fanchin R, Harmas A, Benaoudia F, Lundkvist U, Olivennes F, Frydman R. Microbial flora of the cervix assessed at the time of embryo transfer adversely affects in vitro fertilization outcome. Fertil Steril. 1998 Nov;70(5):866-70. doi: 10.1016/s0015-0282(98)00277-5. PMID 9806568